CLINICAL TRIAL: NCT03542292
Title: Doğumun üçüncü Evresinin yönetiminde Vajinal doğum sonrası Plasental Drenaja karşı Plasenta drenajı: Randomize Bir çalışma
Brief Title: Placental Drainage Versus no Placental Drainage After Vaginal Delivery in the Management of Third Stage of Labour
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeynep Kamil Maternity and Pediatric Research and Training Hospital (Other)
Responsible Party: Principal Investigator, Evrim Bostancı, Principal Investigator, Zeynep Kamil Maternity and Pediatric Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: EY.FR.22
Record Dates: First submitted 2018-05-18; First posted 2018-05-31 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Placental Bleeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placental drainage group (Experimental): In study group; umbilical cord was clamped from fetal side but unclamped from maternal side. After that unclamped side of umblical cord was left open to drain the blood until the flow ceased. The blood was collected in the metal bowl and measured using a measuring jar. Care was taken not to mix the drained blood from the cord with the blood lost during the third stage.
  Interventions: Diagnostic Test: placental drainage
- no placental drainage group (Active Comparator): In control group the umblical cord was clamped both sides.
  Interventions: Diagnostic Test: placental drainage

INTERVENTIONS:
Diagnostic Test: placental drainage

SUMMARY:
In this randomized controlled study, 222 pregnant women who admitted to Zeynep Kamil Women and Children's Health Training and Research Hospital from December 2016 and July 2017 were included. They were randomized into study(111) or control(111) group when they delivered vaginally. In study group; umbilical cord was clamped from fetal side but unclamped from maternal side. After that unclamped side of umblical cord was left open to drain the blood until the flow ceased. In control group the umblical cord was clamped both sides.

DETAILED DESCRIPTION:
This was a randomized controlled trial on 222 pregnant women who admitted to our hospital from December 2016 and July 2017. After approval of the ethics committee and written consent of the patients were taken, 222 pregnant women were included in this study. They were randomized into study(111) or control(111) group when they delivered vaginally. Randomization was performed by means of a computer-generated randomization table.

In study group; umbilical cord was clamped from fetal side but unclamped from maternal side. After that unclamped side of umblical cord was left open to drain the blood until the flow ceased. The blood was collected in the metal bowl and measured using a measuring jar. Care was taken not to mix the drained blood from the cord with the blood lost during the third stage. In control group the umblical cord was clamped both sides.

The inclusion criteria were>37 weeks of gestation, singleton, alive pregnancy, with vertex presentation expected to have spontaneous vaginal delivery. The exclusion criteria were fetal malpresentation, history of postpartum hemorrhage, preterm delivery, multiple pregnancy, fetal anomaly, uterine malformation, fetal demise, women with immediate delivery indications, unable to give written informed consent, a clinically estimated fetal weight >4500, preeclampsia, antepartum hemorrhage, previous cesarean section, instrumental delivery and known coagulation disorders. Patients were recruited regardless of using cervical ripening agents.

General physical and obstetric examination were performed after a detailed history taking. A sample of venous blood was obtained for hemoglobin concentration on admission. Labour was conducted according to the hospital protocol. Labour was augmented with oxytocin in active phase of labour. All patients were monitored with cardiotocography (CTG) before induction of labor and CTG was used continuously during labor. Oxytocin infusion was continued until delivery of both child and placenta, unless complications occurred. For all patients, blood lost in the third stage of labour was measured by collecting the blood in a disposable conical measuring bag. The time of delivery of the neonate was recorded and after then prophylactic uterotonic agents (Synpitan Fort, 5 IU) was given to all patients. Placenta was delivered by controlled cord traction andthe time of placental delivery was noted in both groups. If the placenta had not been delivered spontaneously by 30 minutes after birth, it was removed manually. The vital signs(blood pressure, pulse rate, temperature) uterine tone of the patients were monitored after delivery of neonate and placenta. The hemoglobin concentration was estimated 24 hours after delivery.

The outcome measures were the duration of the third stage of labour, defined as interval from birth of the infant to delivery of the placenta, haemoglobin difference between admission and 24 hours after delivery, visual analog scale (VAS) scores, weight of placenta, need for blood transfusion, blood loss from umbilical cord and blood loss in the third stage of labour. PPH was defined as a loss of more than 500 mL of blood within the first 24 hours following childbirth.

ELIGIBILITY:
Inclusion Criteria:

>37 weeks of gestation, singleton, alive pregnancy, with vertex presentation expected to have spontaneous vaginal delivery -

Exclusion Criteria:

fetal malpresentation, history of postpartum hemorrhage, preterm delivery, multiple pregnancy, fetal anomaly, uterine malformation, fetal demise, women with immediate delivery indications, unable to give written informed consent, a clinically estimated fetal weight >4500, preeclampsia, antepartum hemorrhage, previous cesarean section, instrumental delivery known coagulation disorders.

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 222 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
the duration of the third stage of labour | minutes from baby delivery to delivery of the placenta
  interval from birth of the infant to delivery of the placenta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Asicioglu O, Unal C, Asicioglu BB, Temizkan O, Yildirim G, Arici B, Gulova S. Influence of placental cord drainage in management of the third stage of labor: a multicenter randomized controlled study. Am J Perinatol. 2015 Mar;32(4):343-50. doi: 10.1055/s-0034-1384639. Epub 2014 Aug 11. PMID 25111038
- [Result] Soltani H, Poulose TA, Hutchon DR. Placental cord drainage after vaginal delivery as part of the management of the third stage of labour. Cochrane Database Syst Rev. 2011 Sep 7;2011(9):CD004665. doi: 10.1002/14651858.CD004665.pub3. PMID 21901693
- [Result] Roy P, Sujatha MS, Bhandiwad A, Biswas B, Chatterjee A. Placental Blood Drainage as a Part of Active Management of Third Stage of Labour After Spontaneous Vaginal Delivery. J Obstet Gynaecol India. 2016 Oct;66(Suppl 1):242-5. doi: 10.1007/s13224-016-0857-3. Epub 2016 Mar 12. PMID 27651611